CLINICAL TRIAL: NCT00880581
Title: A Phase 2 Study of Intratumoral Injection PF-3512676 in Combination With Local Radiation in Low-Grade B-Cell Lymphomas
Brief Title: A Phase 2 Intratumoral Injection PF-3512676 Plus Local Radiation in Low-Grade B-Cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ronald Levy (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Ronald Levy, Robert K. and Helen K. Summy Professor in the School of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-14820; SU-03272009-2038 (Other: SU IRB); LYMNHL0064 (Other: OnCore)
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma; Lymphomas: Non-Hodgkin Follicular / Indolent B-Cell; Lymphomas: Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-3512676 (Experimental): Patients will be treated with 18 mg PF-3512676 by intratumoral injection on day 2 following local radiotherapy, then weekly for a total of 10 injections over 10 weeks.
  Interventions: Drug: PF-3512676; Radiation: Local radiotherapy

INTERVENTIONS:
Drug: PF-3512676 — 18 mg injection
  Other Names: CpG 7909; CpG; ProMune
Radiation: Local radiotherapy — 2 gray (2 Gy) on each of Days 1 and 2

SUMMARY:
To assess the feasibility of using intra-tumoral PF-3512676 in combination with local radiation as a therapy for lowgrade b-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed low-grade B-cell lymphoma diagnosed as follicular grade 1 or 2, marginal zone or small lymphocytic lymphoma of any initial stage.
* Patients may be either treatment-naïve; relapsed from; or refractory to prior therapy. (15 treatment-naïve and 15 relapsed/refractory patients will be enrolled)
* Patients must have at least one site of disease that is accessible for intratumoral injection of PF-3512676 percutaneously
* Tumor specimens must be available for immunological studies either from a previous biopsy or a new biopsy obtained before the initiation of the study.
* Patients must have measurable disease other than the injection site or biopsy site.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥ 1
* Karnofsky Performance Status (KPS) of ≥ 70
* ≥ 18 years of age
* White blood cells (WBC) ≥ 2,000/uL
* Platelet count ≥ 75,000/mm³
* Absolute neutrophil count (ANC) ≥ 1000
* Serum creatinine ≤ 2.0 mg/dL.
* Bilirubin ≤ 1.5 mg/dL
* Serum glutamic oxalocetic transaminase (SGOT) / serum glutamic pyruvic transaminase (SGPT) ratio < 3 x upper limit of normal (ULN)
* Required wash out periods for prior therapy:

  * Topical therapy: 2 weeks
  * Chemotherapy: 4 weeks
  * Radiotherapy: 4 weeks
  * Other investigational therapy: 4 weeks
  * Rituximab: 12 weeks
* Patients of reproductive potential and their partners must agree to use an effective (>90% reliability) form of contraception during the study and for 4 weeks following the last study drug administration.
* Women of reproductive potential must have a negative urine pregnancy test.
* Life expectancy > 4 months.
* Able to comply with the treatment schedule.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pre-existing autoimmune or antibody mediated disease including:

  * Systemic lupus, erythematosus
  * Rheumatoid arthritis
  * Multiple sclerosis
  * Sjogren's syndrome
  * Autoimmune thrombocytopenia, but excluding controlled thyroid disease
  * Presence of autoantibodies without clinical autoimmune disease.
* Known history of human immunodeficiency virus (HIV).
* Patients with active infection or with a fever > 38.5 C within 3 days prior to the first scheduled treatment.
* Central nervous system (CNS) metastases
* Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.
* History of allergic reactions attributed to compounds of similar composition to PF-3512676
* Current anticoagulant therapy [aspirin (ASA) ≤ 325 mg per day allowed]
* Significant cardiovascular disease [ie, New York Heart Association (NYHA) class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias].
* Pregnant or lactating.
* Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-3512676: To assess the feasibility of using intra-tumoral PF-3512676 (CpG 7909 or ProMune) at 18 mg per week over 10 weeks in combination with local radiation [2 gray (2Gy) on each of Days 1 and 2] as a therapy for low-grade B-cell lymphoma.
Period: Cycle 1
Arm/Group | PF-3512676
Started | 30
Completed | 30
Not Completed | 0
Period: Cycle 2 Re-treatment
Arm/Group | PF-3512676
Started | 24 (6 subjects with progessive disease were not treated and evaluated in Cycle 2)
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-3512676: To assess the feasibility of using intra-tumoral PF-3512676 in combination with local radiation as a therapy for lowgrade b-cell lymphoma.
Arm/Group | PF-3512676
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall ObjectiveResponse (ORR) Rate
Description: Overall objective response rate (OOR) at time of best response was assessed as the sum of the Complete Response (CR) rate and the Partial Response (CR, PR) rate. Response was assessed per the Cheson Criteria, as below.
  * Complete Response (CR) = Complete disappearance of all lesions, evidence, and effects of disease
  * CR/unconfirmed (CRu) = residual lymph node mass >1.5 cm but regressed >75%, with 1 residual lymph node mass >1.5 cm that has regressed by >75% and/or increased number or size of bone marrow aggregates without cytologic or architectural atypia
  * Partial Response (PR) = ≥50% decrease in SPD of the 6 largest lesions with no increase in the size of the other nodes; splenic / hepatic nodules regress ≥50%, and with no new sites of disease Stable disease (SD) = less than PR.
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- PF-3512676: Patients will be treated with 18 mg PF-3512676 by intratumoral injection on day 2 following local radiotherapy, then weekly for a total of 10 injections over 10 weeks.
  PF-3512676: 18 mg injection
  Local radiotherapy: 2 x 2 Gy
Arm/Group | PF-3512676
Number analyzed (Participants) | 30
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 7
  Stable Disease (SD) | 19
  Progressive Disease (PD) | 4

2. Secondary Outcome: Response Rate After Cycle 2
Description: Response after a second cycle of treatment was assessed per the Cheson Criteria, as below.
  * Complete Response (CR) = Complete disappearance of all lesions, evidence, and effects of disease
  * CR/unconfirmed (CRu) = residual lymph node mass >1.5 cm but regressed >75%, with 1 residual lymph node mass >1.5 cm that has regressed by >75% and/or increased number or size of bone marrow aggregates without cytologic or architectural atypia
  * Partial Response (PR) = ≥50% decrease in SPD of the 6 largest lesions with no increase in the size of the other nodes; splenic / hepatic nodules regress ≥50%, and with no new sites of disease Stable disease (SD) = less than PR.
Time Frame: 6 months
Population: Participants with progressive disease (PD) were not re-evaluated.
Measure: Number; unit: participants
Arm/Group | PF-3512676
Number analyzed (Participants) | 20
participants
  Complete Response (CR) | 2
  Stable Disease (SD) | 14
  Partial Response (PR) | 4

ADVERSE EVENTS:
Arm/Group | PF-3512676
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 22/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-3512676 (N=30)
erythema (Skin and subcutaneous tissue disorders) | 17 (17)
headache (General disorders) | 6 (6)
myalgia (Musculoskeletal and connective tissue disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No